CLINICAL TRIAL: NCT07314710
Title: Factors Affecting Postural Awareness in Academics in Kütahya
Brief Title: Factors Affecting Postural Awareness in Academics
Status: Completed | Type: Observational
Sponsor: Kutahya Health Sciences University (Other)
Responsible Party: Principal Investigator, Lütfiye AKKURT, MSc, Assistant Professor, Kutahya Health Sciences University
Other Study IDs: 2025/11-29
Record Dates: First submitted 2025-12-18; First posted 2026-01-02 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Health Adult Subjects
Keywords: postural awareness; academics; posture

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of the study is to determine the factors affecting postural awareness in academics.

DETAILED DESCRIPTION:
The aim of the study is to determine the factors affecting postural awareness in academics. Data on age, height, weight, body mass index, gender, duration of academic work, daily working time, and distance from the eye to the screen were collected. Postural awareness, mindfulness, fatigue, and posture measures are described below. Postural Awareness Scale, Mindfulness Attention Awareness Scale, Chalder Fatigue Scale and New York Posture Rating scale were used in study.

ELIGIBILITY:
Inclusion Criteria:

* Being an academician
* Being between 24 and 60 years old and People and pregnant women were excluded from the study.

Exclusion Criteria:

* Having with any orthopaedic or neurological disorders
* Being pregnant

Ages: 24 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Academics in Kütahya Health Sciences University
Sampling Method: Probability Sample
Enrollment: 122 (Actual)
Dates: Start 2025-09-01 (Actual); Primary Completion 2025-12-10 (Actual); Study Completion 2025-12-18 (Actual)

PRIMARY OUTCOMES:
Postural Awareness Scale | At the beginning of the study
  The Postural Awareness Scale (PAS) was designed by Cramer et al. 1 to measure self-reported awareness of body posture, and translated to Turkish version by Dursun et al.. The PAS consist of 12 items in original form but 12th item was removed from the Turkish version due to factor load was low. The PAS consist of two factor structures, ease/familiarity with postural awareness (items 6-11) and need for attention regulation with postural awareness (items 1-5). The Turkish version of PAS scores range from 11 to 77, higher scores indicate high greater postural awareness. The total score was calculated after reversing the values of items 1, 2, 3, 4, 5 and adding other items.

SECONDARY OUTCOMES:
Mindfulness Attention Awareness Scale | At the beginning of the study
  The Mindfulness Attention Awareness Scale (MAAS) was developed by Brown and Ryan 3 and translated to Turkish version by Özyeşil et al. The MAAS contains 15 items to measure individual differences in the tendency to be mindful. All the items are scored range from 1 (almost never) to 6 (almost always) points. The MAAS total scores can range from 1 to 6 points due to based on a mean (average) of the 15 items. Higher scores indicate a higher level of mindfulness.
Chalder Fatigue Scale | At the beginning of the study
  The Chalder Fatigue Scale (CFS) was developed by Chalder et al. 5 and translated to Turkish version by Adın et al. The CFS measures the severity of perceived fatigue and chronicity of fatigue. The CFS consist of 11 items, and which consist of two dimensions, including physical (CFS-PF) and mental fatigue (CFS-MF). The total score ranges from 0 to 33 points. Higher scores indicates a high level of fatigue.
New York Posture Rating Scale | At the beginning of the study
  The New York Posture Rating (NYPR) Scale was used to assess postural alignment changes for clinical postural evaluation in 13 body aligment segment. Lateral and posterior posture analysis is performed in 13 regions (head, neck, shoulder, scapula, upper thoracic, waist, rips, abdomen, hips, knees, legs, feet and toes). Every region was scored 1 (pronounced deviation), 3 (slight deviation) or 5 (correct posture) points. Total score is between 13-65 points. Higher scores indicates better the postural alignment.

CONTACTS AND LOCATIONS:
Overall Officials: Lütfiye AKKURT, PhD, Principal Investigator — Kütahya Health Sciences University; Nisa TÜRÜTGEN, MSc, Study Chair — Kütahya Health Sciences University
Locations (1):
- Kütahya Health Sciences University, Kütahya, Kütahya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No